CLINICAL TRIAL: NCT02451176
Title: A Prospective Randomized Trial of Biologic Mesh Versus Synthetic Mesh for the Repair of Complex Ventral Hernias
Brief Title: Biologic Mesh Versus Synthetic Mesh in Repair of Ventral Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Rosen (Other)
Responsible Party: Sponsor-Investigator, Michael Rosen, Michael Rosen, MD, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 14-1571; NCT01746316 (obsolete NCT alias)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator: Davol Bard ®Soft Mesh (Active Comparator): Device: Davol Bard ®Soft Mesh Synthetic mesh for open ventral hernia repair for clean-contaminated or contaminated abdominal wall hernias Other Name: synthetic mesh SoftMesh™ (CR Bard)
  Interventions: Device: Davol Bard Soft Mesh synthetic
- Active Comparator: LifeCell Strattice® (Active Comparator): Device: LifeCell Strattice® Reconstructive Tissue Matrix Biologic mesh for open ventral hernia repair for clean-contaminated or contaminated abdominal wall hernias Other Name: Biologic mesh Strattice
  Interventions: Device: LifeCell Strattice Reconstructive Tissue Biologic

INTERVENTIONS:
Device: Davol Bard Soft Mesh synthetic — soft mesh synthetic
  Arms: Active Comparator: Davol Bard ®Soft Mesh
Device: LifeCell Strattice Reconstructive Tissue Biologic — biologic mesh
  Arms: Active Comparator: LifeCell Strattice®

SUMMARY:
This study will compare the safety, efficacy and cost effectiveness of a permanent synthetic mesh versus a biologic prosthesis for the repair of ventral hernias in the setting of clean-contaminated (Class 2) or contaminated (Class 3) surgical procedures. The findings of this study will have a major impact on the field of hernia surgery as it will provide objective guide to mesh selection, optimize surgical approaches for complex ventral hernia repair, and ultimately significantly improve patient outcomes.

DETAILED DESCRIPTION:
This is a multicenter prospective double-blinded randomized controlled trial comparing 253 patients with clean-contaminated (Class 2)or contaminated (Class3) abdominal wall ventral hernias undergoing single staged repair. Soft Mesh by CR Bard, a macroporous monofilament polypropylene permanent mesh will be compared to Strattice mesh by Lifecell, a non-cross linked porcine dermal biologic graft for the single stage open reconstruction of clean-contaminated and contaminated abdominal wall defects. The primary outcome variable will be the absence of surgical site occurence requiring procedural intervention and the absence of a hernia recurrence from the time of surgery up to 24 months of postoperative follow up.

Patients undergoing open ventral hernia repair for clean-contamination and contaminated abdominal wall hernias meeting inclusion criteria will be randomized to receive a synthetic mesh or a biologic mesh. Randomization will be carried out using computer-generated randomization blocks at the time of enrollment. Stratified randomized will be used with the strata formulated by medical center then by clean-contaminated or contaminated surgical site class. The Investigator will be blinded to patient randomization assignment until the point of intra-operative device use following final CDC wound classification, whereas patients and co-investigators responsible for data analysis will remain blinded to patient randomization until the conclusion of the study period. As such, a double-blinded study protocol will be maintained. Patients randomized to synthetic mesh will receive SoftMesh™ (CR Bard, Murray Hill, NJ) and those patients randomized to biologic mesh will receive Strattice™ (Lifecell, Branchburg NJ). The use of biologic and synthetic mesh in contaminated fields is considered experimental however the selection of these prosthetics was based on a careful review of the multiple animal models, preclinical data, and our own clinical experience with each of these materials placed in both clean and contaminated abdominal wall reconstructions. Surgical wounds will be classified based on CDC(Centers for Disease Control) criteria and only Class 2 and 3 wounds will be included in this study.

Postoperatively patients will be evaluated for signs and symptoms of complications along with presence or absence of Surgical Site Infections per CDC guidelines, presence or absence of surgical site occurrences (SSOs) and any procedural interventions required to treat these SSOs, presence or absence of hernia recurrence and any reoperations, length of hospital stay, discharge date, time to return of bowel function and any readmission.

Active participation in this study will last for 24 months and will involve one preoperative evaluation visit, one operative procedure visit, and 4 follow up visits. Participants will complete two brief survey questionnaires regarding quality of life, activities and pain.

The second outcome will be to demonstrate that a macroporous light-weight polypropylene mesh is more cost effective strategy than a biologic prosthetic in clean-contaminated and contaminated abdominal wall reconstruction

ELIGIBILITY:
Inclusion Criteria:

1. The subject is > 21 years of age (including women of childbearing age)
2. Scheduled to undergo a planned open single stage reconstruction of a contaminated (CDC wound class2 or 3) abdominal wall defect
3. Ability to undergo general anesthesia
4. Is willing and able to give informed consent
5. Is this a clean-contaminated (Class 2) or contaminated (Class 3) case per CDC Guidelines?
6. Has an estimated parastomal hernia or midline defect size of >9 cm 2 contaminated (CDC wound class 2 or 3) abdominal wall defect by physical /or radiological exam.
7. Can achieve midline fascial closure?
8. Is subject willing to return for scheduled and required study visits? -

Exclusion Criteria:

1. Patients have a defect that the surgeon cannot achieve primary fascial apposition and requires a bridge of mesh.
2. Is the patients BMI over 45 kg/m2?
3. Is the patient currently pregnant?
4. Will undergo a laparoscopic or robotic hernia repair.
5. Do they have a class 1 or 4 wound per CDC Guidelines?
6. Are they on immunosuppression including medically-induced with>10 mg of prednisone/day?
7. Do they have a collagen vascular disorder?
8. Is patient having a prior mesh removed due to a current active mesh infection? (A synthetic mesh that is not incorporated into the tissue, is extracorporeally exposed or has a chronic draining sinus with clear fluid around the material, but not including synthetic mesh incorporated in abdominal wall and not infected)
9. Does the patient have Ascites refractory to medical management?
10. Are they in end stage renal (on hemodialysis or peritoneal dialysis) or pre-existing liver disease (Hepatitis B or C or Total Bilirubin >3.0mg/dl)?
11. Is the patient severely malnourished as defined by serum albumin<2.0g/dl?
12. Do they have a smoking history within 1 month of surgery?
13. Does the patient have an objection to the implantation of porcine products?
14. Is the subject participating in another clinical study?
15. Are unable to undergo successful retro-rectus/preperitoneal mesh placement

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-04; Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosen, MD, Principal Investigator — Cleveland Clinic, Cleveland, Ohio, United States, 44195
Locations (4):
- United States (4):
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - University of South Carolina School of Medicine, Greenville, South Carolina
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Miller BT, Krpata DM, Petro CC, Beffa LRA, Carbonell AM, Warren JA, Poulose BK, Tu C, Prabhu AS, Rosen MJ. Biologic vs Synthetic Mesh for Parastomal Hernia Repair: Post Hoc Analysis of a Multicenter Randomized Controlled Trial. J Am Coll Surg. 2022 Sep 1;235(3):401-409. doi: 10.1097/XCS.0000000000000275. Epub 2022 Aug 10. PMID 35588504
- [Derived] Rosen MJ, Krpata DM, Petro CC, Carbonell A, Warren J, Poulose BK, Costanzo A, Tu C, Blatnik J, Prabhu AS. Biologic vs Synthetic Mesh for Single-stage Repair of Contaminated Ventral Hernias: A Randomized Clinical Trial. JAMA Surg. 2022 Apr 1;157(4):293-301. doi: 10.1001/jamasurg.2021.6902. PMID 35044431

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Comparator: Davol Bard ®Soft Mesh | Active Comparator: LifeCell Strattice®
Started | 126 | 127
Completed | 126 | 127
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Davol Bard ®Soft Mesh | Active Comparator: LifeCell Strattice® | Total
Number analyzed (Participants) | 126 | 127 | 253
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 63.7 [55 to 69.4] | 63.7 [55.5 to 70.2] | 63.7 [55.4 to 70.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 71 | 136
  Male | 61 | 56 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian not Hispanic | 116 | 115 | 231
  Hispanic | 2 | 0 | 2
  African American | 7 | 12 | 19
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Surgical Site Occurrence Requiring Procedural Intervention
Time Frame: 2 years from surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Davol Bard ®Soft Mesh | Active Comparator: LifeCell Strattice®
Number analyzed (Participants) | 126 | 127
Participants
  No surgical site occurrence requiring procedural intervention | 124 | 126
  Presence of surgical site occurrence requiring procedural intervention | 2 | 1

2. Primary Outcome: Total Number of Participants With Recurrence of Hernias
Time Frame: 2 years post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Davol Bard ®Soft Mesh | Active Comparator: LifeCell Strattice®
Number analyzed (Participants) | 115 | 118
Participants | 7 | 24

3. Secondary Outcome: Direct Costs Associated With the Use of Either Polypropylene or Biologic Mesh
Description: Calculate and compare incremental cost effectiveness ratios for patients undergoing repair of clean-contaminated or contaminated ventral hernias using either polypropylene mesh or biologic mesh
Time Frame: 30 days post surgery
Measure: Median (Inter-Quartile Range); unit: US Dollars
Arm/Group | Active Comparator: Davol Bard ®Soft Mesh | Active Comparator: LifeCell Strattice®
Number analyzed (Participants) | 105 | 103
US Dollars
  Direct cost Surgical Admission | 17110 [14044 to 22677] | 44530 [35172 to 52496]
  Total 30 day direct cost | 17289 [14643 to 23901] | 44936 [35887 to 54656]

ADVERSE EVENTS:
Time Frame: 2 years post surgery
Arm/Group | Active Comparator: Davol Bard ®Soft Mesh | Active Comparator: LifeCell Strattice®
All-Cause Mortality (participants affected / at risk) | 5/126 | 6/127
Serious Adverse Events (participants affected / at risk) | 11/126 | 11/127
Other Adverse Events (participants affected / at risk) | 108/126 | 103/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Davol Bard ®Soft Mesh (N=126) | Active Comparator: LifeCell Strattice® (N=127)
Surgical Site Infection (Infections and infestations) | 4 (4) | 3 (3)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Non-Healing wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 1 (1) | 0 (0)
Foreign Body Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Obstruction of Transplant Ureter (Product Issues) | 1 (1) | 0 (0)
Mesh Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Bowel Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seroma (General disorders) | 0 (0) | 1 (1)
nsertion of Peripheral Central Venous Access Device (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Davol Bard ®Soft Mesh (N=126) | Active Comparator: LifeCell Strattice® (N=127)
Surgical Site Infection (Infections and infestations) | 9 (9) | 17 (17)
Esophageal Stricture (Gastrointestinal disorders) | 0 (0) | 1 (10)
Esophageal Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (10)
Ileus (Gastrointestinal disorders) | 21 (21) | 18 (18)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 6 (6)
Pouchitis (Infections and infestations) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Wound Infection (Infections and infestations) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Bowel Obstruction (Gastrointestinal disorders) | 9 (9) | 3 (3)
Seroma (General disorders) | 4 (4) | 4 (4)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 7 (7) | 12 (12)
C-Diff (Infections and infestations) | 3 (3) | 2 (2)
Suture Abscess (Infections and infestations) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Incisional Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Organ Space Infection (Infections and infestations) | 2 (2) | 0 (0)
Non-Healing Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Dehydration (General disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 4 (4)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
PICC line infection (Infections and infestations) | 0 (0) | 1 (1)
Urine Leak (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Scar Revision (Surgical and medical procedures) | 1 (1) | 0 (0)
Drainage for JP removal site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Torn Retina (Eye disorders) | 1 (1) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Upper Lip Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Bowel Enterotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT02451176/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT02451176/ICF_001.pdf